CLINICAL TRIAL: NCT02602405
Title: Return to Work After Potential Severe Injury; a Population Based Observational Study
Brief Title: Return to Work After Potential Severe Injury
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Statistics Norway (Industry); Namsos Hospital (Other); Helse Nord-Trøndelag HF (Other); Alesund Hospital (Other); Molde Hospital (Other); Kristiansund Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/1582
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Multiple Trauma
Keywords: Outcome Assessment (Health Care); Return to work; Registries; Norway
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Norway an estimated 10 % of the population is injured annually. Of these 36.000 sustain permanent functional impairment, 1.200 receive disability pension, and approximately 2.500 die because of their injuries. Mortality is the most common variable measuring trauma outcome. However, measuring only trauma mortality may be looking merely at the tip of the iceberg. For every trauma death, there are ten-folds suffering long term functional impairment. Mortality is therefore a too crude variable to describe the impact of injuries - both for the individual trauma patient and for society as a whole. There is a need for variables describing long-term outcomes on a functional level. The aim of this study is to use the rate of return to work and education as an alternative outcome measure. The ability of returning to work after injury is a central indicator of individual functional outcome, combining both physical and mental skills in performing complex and compound tasks. Previous studies on return to work after injury are limited by a combination of short follow-up times, the use of patient reported outcomes and having mainly been focusing on only severely injured patients (ISS > 15). This a population-based study including all patients in working age (16 - 65 years) received by a trauma team in any of the eight hospitals within the region of Central Norway in the time period from June 1st,2007 to May 30th, 2010. Already collected trauma registry data will be linked with national register data on sickness and disability benefits, employment and education.

ELIGIBILITY:
Inclusion Criteria:

* exposed to traumatic injuries
* received by trauma team attendance
* received by trauma team activation protocol

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in working age received by a trauma team in any of the eight hospitals within the region of Central Norway in the period from June 1st, 2007 to May 30th, 2010
Sampling Method: Non-Probability Sample
Enrollment: 1741 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Return to work | up to 8 years
Return to education | up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Pål Klepstad, md prof, Study Director — Norwegian University of Science and Technology
Locations (8):
- Norway (8):
  - Ålesund Hospital, Ålesund
  - Kristiansund Hospital, Kristiansund
  - Levanger Hospital, Levanger
  - Molde Hospital, Molde
  - Namsos Hospital, Namsos
  - Orkanger Hospital, Orkanger
  - St Olavs Hospital, Trondheim
  - Volda Hospital, Volda

REFERENCES:
- [Derived] Uleberg O, Pape K, Kristiansen T, Romundstad PR, Klepstad P. Population-based analysis of the impact of trauma on longer-term functional outcomes. Br J Surg. 2019 Jan;106(1):65-73. doi: 10.1002/bjs.10965. Epub 2018 Sep 17. PMID 30221344